CLINICAL TRIAL: NCT07263763
Title: Clinical and Microbiological Characteristics of Orthodontic Patients With Fixed Appliances Treated for Gingival Hyperplasia Using Surgical Scalpel and Diode Laser: A Randomized Clinical Trial.
Brief Title: Gingival Hyperplasia Treatment With Surgical Scalpel vs Diode Laser in Orthodontic Patients.
Acronym: GINGILASCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Thu Thuy (Other)
Responsible Party: Sponsor-Investigator, Nguyen Thu Thuy, Associate Professor - PhD, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1427/ĐHYD-HDDD; 1427/ĐHYD-HĐĐĐ (Other: University of Medicine and Pharmacy at Ho Chi Minh City)
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Gingival Enlargement
Keywords: Gingival overgrowth; Gingival enlargement; Orthodontic treatment; Laser gingivectomy; Surgical gingivectomy; Diode laser; Fixed orthodontic appliances; Randomized clinical trial
MeSH Terms: conditions — Gingival Hyperplasia; Gingival Overgrowth

STUDY DESIGN:
Intervention Model Description: This is a randomized, split-mouth clinical trial using a crossover design. Each participant received both interventions (scalpel gingivectomy and diode laser gingivectomy) at different sites within the same arch.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions, masking of participants and operators was not feasible. Outcome assessors were blinded to the type of intervention performed at each site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalpel Gingivectomy (Experimental): Conventional gingivectomy performed using a surgical scalpel. Gingival overgrowth was excised using standard surgical technique under local anesthesia.
  Interventions: Procedure: Scalpel Gingivectomy
- Diode Laser Gingivectomy (Experimental): Gingivectomy performed using a diode laser. Laser parameters were set according to manufacturer's recommendations. No sutures required.
  Interventions: Procedure: Diode laser Gingivectomy

INTERVENTIONS:
Procedure: Scalpel Gingivectomy — Conventional gingivectomy performed using a surgical scalpel. Gingival overgrowth was excised using standard surgical technique under local anesthesia.
  Arms: Scalpel Gingivectomy
Procedure: Diode laser Gingivectomy — Gingivectomy performed using a diode laser. Laser parameters were set according to manufacturer's recommendations. No sutures required.
  Arms: Diode Laser Gingivectomy

SUMMARY:
Gingival enlargement is a common complication in orthodontic patients, often resulting from plaque accumulation and chronic inflammatory response during fixed appliance therapy. Surgical gingivectomy is frequently required to restore gingival contour, improve esthetics, and facilitate oral hygiene. Traditionally, gingivectomy is performed using a scalpel, but laser-assisted techniques have recently gained popularity due to their potential benefits, including reduced bleeding, postoperative discomfort, and faster healing.

This randomized split-mouth clinical trial aims to compare the clinical and microbiological outcomes of gingivectomy performed with a diode laser versus conventional scalpel surgery in orthodontic patients presenting with gingival enlargement. Clinical parameters, microbial profiles, and patient-reported outcomes will be evaluated at baseline and at multiple postoperative intervals to assess the effectiveness and advantages of each technique.

DETAILED DESCRIPTION:
Gingival enlargement is a frequent periodontal manifestation in patients undergoing fixed orthodontic treatment, primarily resulting from increased plaque retention and subsequent chronic inflammation. This condition can compromise esthetics, interfere with effective oral hygiene, and lead to periodontal complications if left untreated. Gingivectomy is the treatment of choice for removing excess gingival tissue and reestablishing physiological gingival contours. Conventional scalpel gingivectomy has been widely used; however, the advent of laser technology, particularly diode lasers, has provided an alternative surgical approach with potential clinical advantages, including better hemostasis, reduced intraoperative discomfort, faster wound healing, and less postoperative pain.

This study is designed as a randomized split-mouth clinical trial to compare the clinical and microbiological outcomes of gingivectomy performed using a scalpel versus a diode laser in orthodontic patients with gingival enlargement. Eligible participants will be recruited from the Orthodontics Department of the Ho Chi Minh City National Hospital of Odonto-Stomatology. Each patient will undergo gingivectomy on two contralateral quadrants: one quadrant treated with conventional scalpel surgery (control side) and the other with diode laser surgery (test side). The allocation of quadrants will be randomized.

Clinical parameters including Plaque Index (PlI), Gingival Index (GI), Probing Pocket Depth (PPD), Gingival Margin Position (GMP), and Bleeding on Probing (BoP) will be recorded at baseline and at multiple postoperative intervals. Subgingival plaque samples will be collected for microbiological analysis using real-time polymerase chain reaction (qPCR) to evaluate the presence and levels of periodontopathogenic bacteria. Patient-reported outcomes such as postoperative pain will also be assessed using a visual analog scale (VAS).

All surgical procedures will be performed by the same calibrated operator to minimize variability. Standardized oral hygiene instructions will be provided to all participants throughout the study period. The collected data will be analyzed to determine differences in clinical healing, microbial changes, and patient comfort between the two treatment modalities. The findings are expected to provide evidence-based insights into the advantages and limitations of diode laser gingivectomy compared with the traditional scalpel technique in orthodontic patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older who agree to take part in the study.
* Individuals in good general health with no history of systemic diseases.
* Patients undergoing fixed orthodontic treatment with metallic brackets for at least 6 months and presenting with gingival enlargement.
* Patients with good oral hygiene (Plaque Index [PlI] < 1) and who comply with the instructions provided by the dentist during the treatment period.

Exclusion Criteria:

* History of using medications associated with gingival enlargement, such as anticonvulsants, immunosuppressants, or calcium channel blockers (e.g., phenytoin, cyclosporine, nifedipine, verapamil, diltiazem, felodipine, nitredipine, etc.).
* Pregnant or breastfeeding women, or individuals using hormonal therapy.
* Patients who have undergone periodontal treatment within the last 6 months.
* Use of antibiotics within 3 months prior to study enrollment.
* Presence or history of systemic diseases.
* Patients who refuse the use of laser in treatment.
* Patients who are uncooperative, have poor oral hygiene (PlI > 1), discontinue participation during the study, or fail to follow instructions throughout the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Gingival margin position | 1 month and 3 months after gingivectomy
  Reduction in Gingival Overgrowth Index

SECONDARY OUTCOMES:
Probing Pocket Depth (PPD) Reduction | 1 month and 3 months after gingivectomy
  Changes in probing pocket depth at baseline and follow-up to assess periodontal healing response.
Reduction in Gingival Index (GI) | 1 month and 3 months after gingivectomy
  Changes in gingival inflammation as assessed by the Löe and Silness Gingival Index at baseline, 1 month and 3 months after treatment.
Reduction in Plaque Index (PlI) | 1 month and 3 months after gingivectomy
  Changes in plaque accumulation as measured by the Silness and Löe Plaque Index at baseline, 1 month and 3 months post-treatment.
Reduction in Bleeding on Probing (BoP) | 1 month and 3 months after gingivectomy
  Changes in bleeding on probing percentage recorded at baseline, 1 month and 3 months after treatment to evaluate periodontal health response.
Microbiological changes in subgingival plaque | 1 month and 3 months after gingivectomy
  hanges in subgingival bacterial composition (e.g., total bacterial load, presence of periodontal pathogens) between baseline, 1 month and 3 months after treatment.
Postoperative pain score | 1 day, 3 days and 7 days after gingivectomy
  Patient-reported pain intensity measured using the Visual Analog Scale (VAS) to compare postoperative discomfort between treatment groups.
Post-surgical bleeding | 1 day, 3 days and 7 days post-surgery
  Assessment of postoperative bleeding severity and duration based on clinical observation and patient reports, to compare healing response between scalpel and diode laser techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Thi Hong Nhung Nguyen, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City - Faculty of Odonto-Stomatology, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared because the study is conducted as part of a postgraduate thesis with a limited scope and without a formal data sharing agreement.

REFERENCES:
- [Result] Newman MG, Takei H, Klokkevold PR, Carranza FA. Newman and Carranza's Clinical Periodontology and Implantology. 14th ed. St. Louis: Elsevier / Saunders; 2023.
- [Result] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Result] Krishnan V, Ambili R, Davidovitch Z, Murphy NC. Gingiva and Orthodontic Treatment. Semin Orthod. 2007;13(4):257-271. doi:10.1053/j.sodo.2007.08.007.
- [Result] Fornaini C, Rocca JP, Bertrand MF, Merigo E, Nammour S, Vescovi P. Nd:YAG and diode laser in the surgical management of soft tissues related to orthodontic treatment. Photomed Laser Surg. 2007 Oct;25(5):381-92. doi: 10.1089/pho.2006.2068. PMID 17975951
- [Result] Maboudi A, Fekrazad R, Shiva A, Salehabadi N, Moosazadeh M, Ehsani H, Yazdani O. Gingivectomy with Diode Laser Versus the Conventional Scalpel Surgery and Nonsurgical Periodontal Therapy in Treatment of Orthodontic Treatment-Induced Gingival Enlargement: A Systematic Review. Photobiomodul Photomed Laser Surg. 2023 Sep;41(9):449-459. doi: 10.1089/photob.2023.0060. PMID 37738371
- [Result] Lione R, Pavoni C, Noviello A, Clementini M, Danesi C, Cozza P. Conventional versus laser gingivectomy in the management of gingival enlargement during orthodontic treatment: a randomized controlled trial. Eur J Orthod. 2020 Jan 27;42(1):78-85. doi: 10.1093/ejo/cjz032. PMID 31111882
- [Result] Zanatta FB, Ardenghi TM, Antoniazzi RP, Pinto TM, Rosing CK. Association between gingival bleeding and gingival enlargement and oral health-related quality of life (OHRQoL) of subjects under fixed orthodontic treatment: a cross-sectional study. BMC Oral Health. 2012 Nov 27;12:53. doi: 10.1186/1472-6831-12-53. PMID 23186371
- [Result] Gong Y, Lu J, Ding X. Clinical, microbiologic, and immunologic factors of orthodontic treatment-induced gingival enlargement. Am J Orthod Dentofacial Orthop. 2011 Jul;140(1):58-64. doi: 10.1016/j.ajodo.2010.02.033. PMID 21724088
- See also: University of Medicine and Pharmacy at Ho Chi Minh City — https://ump.edu.vn